CLINICAL TRIAL: NCT02432430
Title: Comparison of Immunization Quality Improvement Dissemination Study
Acronym: CIzQIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Linda Fu, Associate Professor of Pediatrics, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ChildrensRI
Record Dates: First submitted 2015-04-22; First posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Immunization; DTaP Vaccine; Hepatitis B Vaccine; MMR Vaccine; HIB-vaccine; Poliovirus Vaccine, Inactivated; Chickenpox Vaccine; Pneumococcal Polysaccharide Vaccine
Keywords: N05.300.150.410; practice guideline; D20.215.894.899.290.130; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Hepatitis B; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- quality improvement technical support (Experimental): QI support to improve DTP/Hep B/MMR/Var/PCV/Hib/IPV coverage. Participants receive a Vaccinator Toolkit and attend 6 virtual QI Learning Sessions and 12 monthly conference calls with a coach and other participant teams. On a monthly basis for 11 months, participants collect, submit and review immunization data of 10-20 of their patients ages 3 months to 18 months. After 12 months, participants attend a virtual QI Debriefing Session.
  Interventions: Behavioral: QI support to improve DTP/Hep B/MMR/Var/PCV/Hib/IPV coverage
- pay for performance (Active Comparator): Incentives to improve DTP/HepB/MMR/Var/PCV/Hib/IPV coverage. Participants receive a Vaccinator Toolkit and are informed of a tiered incentives structure. Practices receive bonuses for both improvement in individual practice coverage as well as improvement in coverage for all practices allocated to this study arm.
  Interventions: Behavioral: Incentives to improve DTP/HepB/MMR/Var/PCV/Hib/IPV coverage

INTERVENTIONS:
Behavioral: QI support to improve DTP/Hep B/MMR/Var/PCV/Hib/IPV coverage — Quality improvement technical support to help providers' ability to institute best practices to improve delivery of the following vaccines: DTP, HepB, MMR, Var, PCV, Hib, IPV
  Arms: quality improvement technical support
Behavioral: Incentives to improve DTP/HepB/MMR/Var/PCV/Hib/IPV coverage — Financial incentives to support to help providers' ability to institute best practices to improve delivery of the following vaccines: DTP, HepB, MMR, Var, PCV, Hib, IPV
  Arms: pay for performance

SUMMARY:
Dissemination research examines the processes and factors that lead to widespread use of evidence-based interventions. There are several theories on how to best minimize the perceived and actual burdens on practitioners associated with implementing evidence-based medicine. For instance, the pay for performance model attempts to improve physician compliance with quality guidelines by providing financial incentives. Recent studies suggest pay for performance is effective in improving practitioner performance, but it is unclear whether the gains are sustainable once incentives are stopped.

Another approach to promoting best practices is the Model for Improvement whose main method is to employ Plan-Do-Study-Act (PDSA) cycles of small changes Although this approach has been successful within individual institutions, there is minimal evidence of its effect when employed simultaneously in multiple autonomous institutions. There is also little evidence of the sustainability of outcomes after intervention activities end.

The specific aims of the proposed study are to examine the effect of quality improvement dissemination models on the immunization coverage of children ages 3 to 18 months old. The investigators propose to:

1. Determine the effect on immunization compliance of two different models of dissemination which will provide physicians 12 months of quality improvement (QI) activity support for implementing CDC immunization best practices.

Hypothesis 1a: Study participants receiving the QI technical support intervention (QITS) will have more improvement in immunization rates from baseline to immediately after support ends than participants receiving the pay for performance intervention (P4P).

Hypothesis 1b: Study participants receiving QITS will increase immunization coverage for their practices over baseline.

Hypothesis 1c: Study participants receiving P4P will increase immunization coverage for their practices over baseline.

ELIGIBILITY:
Inclusion Criteria:

* regular patient of a participating practice

Exclusion Criteria:

* fewer than 2 encounters at a participating practice
* moved or gone elsewhere prior to assessment date
* medical contraindication to vaccination

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2186 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
relative risk of child being up to date with all age-appropriate vaccines as assessed by random selection of 50 patients per practice for compliance with HepB, DTaP, Hib, PCV, IPV, MMR, Var | 12 months
  receipt of all age-appropriate immunization

SECONDARY OUTCOMES:
percent of all age-appropriate, indicated vaccines received (HepB, DTaP, Hib, PCV, IPV, MMR, Var) | 12 months
  percent of all needed vaccines received

REFERENCES:
- [Derived] Fu LY, Zook K, Gingold JA, Gillespie CW, Briccetti C, Cora-Bramble D, Joseph JG, Haimowitz R, Moon RY. Strategies for Improving Vaccine Delivery: A Cluster-Randomized Trial. Pediatrics. 2016 Jun;137(6):e20154603. doi: 10.1542/peds.2015-4603. Epub 2016 May 10. PMID 27244859